CLINICAL TRIAL: NCT01627756
Title: Continued Mechanical Ventilation During CABG Operation Attenuates Systemic Immune Modulation
Brief Title: Continued Ventilation During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Hendrik Jan Ankersmit, Assoc. Prof, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2894-2008
Record Dates: First submitted 2012-06-19; First posted 2012-06-26 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
Keywords: Thoracic Surgery; Endotoxins; Respiration, Artificial; Immune System
MeSH Terms: conditions — Coronary Artery Disease; Respiratory Aspiration | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventilation Group (Experimental): Volume controlled ventilation was done during the whole surgery.
  Interventions: Other: Lung Ventilation
- Non-ventilation Group (Active Comparator): In the non-ventilated group lungs were collapsed after completion of CPB until after weaning from the extracorporeal circulation.
  Interventions: Other: Non-ventilated Group

INTERVENTIONS:
Other: Lung Ventilation — In the ventilated group, mechanical ventilation was done with the half of the initial tidal volume (i.e. 3-4 ml/kg, 250-300ml) during the aortic cross-clamp.
  Arms: Ventilation Group
Other: Non-ventilated Group — . In the non-ventilated group lungs were collapsed after completion of CPB until after weaning from the extracorporeal circulation.
  Arms: Non-ventilation Group

SUMMARY:
Cardiopulmonary bypass (CPB) is well known to induce a strong anti-inflammatory response. The investigators examined whether continued mechanical ventilation during CPB alters systemic immune activation.

DETAILED DESCRIPTION:
Cardiopulmonary bypass is well known to induce a strong anti-inflammatory response. Studies had been shown that the contact of blood components with artificial surfaces, the surgical trauma, endotoxemia and a reperfusion injury are in part responsible for the seen immunological affect after surgery. The purpose of this study is to test the effect of continued mechanical ventilation during surgery on a blood marker called soluble ST2 in patients sera. Soluble ST2 acts as a decoy receptor of IL-33 and has anti-inflammatory effects. Elevated soluble ST2 concentrations are reported in patients with acute myocardial infarction, sepsis, congestive heart failure and elevates soluble ST2 levels are associated with adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* age > 40 and < 80

Exclusion Criteria:

* treatment with steroids or immunomodulatory interventions during the past four weeks
* signs of an acute infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Alteration of soluble ST2 concentration in serum | Preoperative, postoperative, day 1, day 2, day 3, day 4, day 5 after surgery
  Concentration of soluble ST2 will be assessed in the serum of patient´s preoperativem, postoperative and the following five consecutive days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Jan Ankersmit, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Debrecen, Debrecen, Hungary

REFERENCES:
- [Background] Szerafin T, Niederpold T, Mangold A, Hoetzenecker K, Hacker S, Roth G, Lichtenauer M, Dworschak M, Wolner E, Ankersmit HJ. Secretion of soluble ST2 - possible explanation for systemic immunosuppression after heart surgery. Thorac Cardiovasc Surg. 2009 Feb;57(1):25-9. doi: 10.1055/s-2008-1039044. Epub 2009 Jan 23. PMID 19169993
- [Background] Szerafin T, Hoetzenecker K, Hacker S, Horvath A, Pollreisz A, Arpad P, Mangold A, Wliszczak T, Dworschak M, Seitelberger R, Wolner E, Ankersmit HJ. Heat shock proteins 27, 60, 70, 90alpha, and 20S proteasome in on-pump versus off-pump coronary artery bypass graft patients. Ann Thorac Surg. 2008 Jan;85(1):80-7. doi: 10.1016/j.athoracsur.2007.06.049. PMID 18154785
- [Background] Szerafin T, Horvath A, Moser B, Hacker S, Hoetzenecker K, Steinlechner B, Brunner M, Roth G, Boltz-Nitulescu G, Peterffy A, Wolner E, Ankersmit HJ. Apoptosis-specific activation markers in on- versus off-pump coronary artery bypass graft (CABG) patients. Clin Lab. 2006;52(5-6):255-61. PMID 16812952
- [Background] Szerafin T, Brunner M, Horvath A, Szentgyorgyi L, Moser B, Boltz-Nitulescu G, Peterffy A, Hoetzenecker K, Steinlechner B, Wolner E, Ankersmit HJ. Soluble ST2 protein in cardiac surgery: a possible negative feedback loop to prevent uncontrolled inflammatory reactions. Clin Lab. 2005;51(11-12):657-63. PMID 16329625
- [Background] Mildner M, Storka A, Lichtenauer M, Mlitz V, Ghannadan M, Hoetzenecker K, Nickl S, Dome B, Tschachler E, Ankersmit HJ. Primary sources and immunological prerequisites for sST2 secretion in humans. Cardiovasc Res. 2010 Sep 1;87(4):769-77. doi: 10.1093/cvr/cvq104. Epub 2010 Apr 2. PMID 20363761
- [Background] Ng CS, Arifi AA, Wan S, Ho AM, Wan IY, Wong EM, Yim AP. Ventilation during cardiopulmonary bypass: impact on cytokine response and cardiopulmonary function. Ann Thorac Surg. 2008 Jan;85(1):154-62. doi: 10.1016/j.athoracsur.2007.07.068. PMID 18154801
- [Derived] Beer L, Szerafin T, Mitterbauer A, Debreceni T, Maros T, Dworschak M, Roth GA, Ankersmit HJ. Low tidal volume ventilation during cardiopulmonary bypass reduces postoperative chemokine serum concentrations. Thorac Cardiovasc Surg. 2014 Dec;62(8):677-82. doi: 10.1055/s-0034-1387824. Epub 2014 Dec 15. PMID 25226360
- [Derived] Beer L, Szerafin T, Mitterbauer A, Kasiri MM, Debreceni T Palotas L, Dworschak M, Roth GA, Ankersmit HJ. Ventilation during cardiopulmonary bypass: impact on heat shock protein release. J Cardiovasc Surg (Torino). 2014 Dec;55(6):849-56. Epub 2013 Dec 17. PMID 24343370